CLINICAL TRIAL: NCT01282008
Title: Message Testing for Tobacco-Related Corrective Statements
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911067; 11-C-N067
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2019-01-22

CONDITIONS: Tobacco; Smoking; Communication
Keywords: Online Surveys; Tobacco Corrective Statements; Message Testing; Focus Groups
MeSH Terms: conditions — Smoking; Communication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Focus Groups: Focus Groups about smoking messages

SUMMARY:
BACKGROUND:

This document outlines the study design and procedures to be used to evaluate a series of corrective statements to augment consumer knowledge and beliefs about smoking as related to past actions of tobacco companies. The statements were ordered by a U.S. Federal Court in U.S. v. Philip Morris USA, Inc., and are intended to target potential misperceptions resultant of past marketing and promotion practices undertaken by the tobacco industry.

OBJECTIVES:

The U.S. Department of Justice has asked NCI to take the lead on developing and testing corrective statements with adult and youth audiences to ensure both message comprehension and avoidance of unintended consequences of message exposure, such as boomerang effects, smoking triggers, or knowledge gaps.

The court has identified five areas that the statements shall address:

1. The adverse health effects of smoking;
2. The addictiveness of smoking and nicotine;
3. The lack of any significant health benefit from smoking low tar, light, ultra light, mild, and natural cigarettes;
4. The tobacco industry s manipulation of cigarette design and composition to ensure optimum nicotine delivery;
5. The adverse health effects of secondhand smoke.

ELIGIBILITY:

Message testing will be undertaken with the following audiences:

* Current smokers (with an oversample of low socioeconomic status individuals)
* General population nonsmokers and former smokers (with an oversample of low socioeconomic status individuals)
* Spanish-speaking Hispanics
* Youth age 14-17

DESIGN:

Both qualitative and quantitative methods (focus groups and post-test comparison group Web-enabled surveys) will be used to develop and test a range of corrective statements in the five areas outlined by the court.

* Focus group participants: 48-64
* Survey participants: 2500

DETAILED DESCRIPTION:
BACKGROUND:

This document outlines the study design and procedures to be used to evaluate a series of corrective statements to augment consumer knowledge and beliefs about smoking as related to past actions of tobacco companies. The statements were ordered by a U.S. Federal Court in U.S. v. Philip Morris USA, Inc., and are intended to target potential misperceptions resultant of past marketing and promotion practices undertaken by the tobacco industry.

OBJECTIVES:

The U.S. Department of Justice has asked NCI to take the lead on developing and testing corrective statements with adult and youth audiences to ensure both message comprehension and avoidance of unintended consequences of message exposure, such as boomerang effects, smoking triggers, or knowledge gaps.

The court has identified five areas that the statements shall address:

1. The adverse health effects of smoking;
2. The addictiveness of smoking and nicotine;
3. The lack of any significant health benefit from smoking low tar, light, ultra light, mild, and natural cigarettes;
4. The tobacco industry s manipulation of cigarette design and composition to ensure optimum nicotine delivery;
5. The adverse health effects of secondhand smoke.

ELIGIBILITY:

Message testing will be undertaken with the following audiences:

* Current smokers (with an oversample of low socioeconomic status individuals)
* General population nonsmokers and former smokers (with an oversample of low socioeconomic status individuals)
* Spanish-speaking Hispanics
* Youth age 14-17

DESIGN:

Both qualitative and quantitative methods (focus groups and post-test comparison group Web-enabled surveys) will be used to develop and test a range of corrective statements in the five areas outlined by the court.

* Focus group participants: 48-64
* Survey participants: 2500

ELIGIBILITY:
* INCLUSION CRITERIA:
* Youth age 14-17
* Youth current smokers, former smokers, and never smokers
* Youth male and female genders
* Youth of all race/ethnicity categories, including: White, Black/African American, Asian, Hispanic/Latino, American Indian/Alaskan Native, Native Hawaiian/Pacific Islander

EXCLUSION CRITERIA:

Participants will be excluded from focus groups and survey if they work in:

* Media
* Advertising, market research
* Public health or health promotion
* An employee of the Federal Govemment who works at HHS or DoJ
* The tobacco or alcohol industries

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Random sample of GfK Web panel participants.@@@@@@
Sampling Method: Probability Sample
Enrollment: 627 (Actual)
Dates: Start 2011-01-21

PRIMARY OUTCOMES:
Knowledge | Immediately upon exposure to stimuli
  Tobacco-related knowledge, attitudes, and beliefs were measured at baseline and after exposure to message stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly D Blake, D.Sc., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ayanian JZ, Cleary PD. Perceived risks of heart disease and cancer among cigarette smokers. JAMA. 1999 Mar 17;281(11):1019-21. doi: 10.1001/jama.281.11.1019. PMID 10086437
- [Background] Evans WD, Crankshaw E, Nimsch C, Morgan-Lopez A, Farrelly MC, Allen J. Media and secondhand smoke exposure: results from a national survey. Am J Health Behav. 2006 Jan-Feb;30(1):62-71. doi: 10.5555/ajhb.2006.30.1.62. PMID 16430321
- [Background] Stryker JE, Moriarty CM, Jensen JD. Effects of newspaper coverage on public knowledge about modifiable cancer risks. Health Commun. 2008 Jul;23(4):380-90. doi: 10.1080/10410230802229894. PMID 18702002